CLINICAL TRIAL: NCT07394751
Title: Clinical Performance of Bioactive Restorative Materials in Occlusal Restorations: Preliminary Results of a Split-mouth Study
Brief Title: Clinical Performance of Bioactive Restorative Materials
Acronym: Bioactive
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sebnem Turkun, Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-68869993-000-1477638; 224S847 (Other Grant/Funding Number: Tübitak)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Dental Caries; Dental Adhesive Materials
Keywords: Bioactive Restorative Materials; Dental Restorations; Clinical trial; FDI-2 criteria
MeSH Terms: conditions — Dental Caries | interventions — ACTIVA BioACTIVE-RESTORATIVE

STUDY DESIGN:
Intervention Model Description: Randomized split mouth study design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tetric N-Ceram BulkFill (Active Comparator): Tetric N-Ceram Bulkfill application (control group; device 1) was randomly applied to patients.
  Interventions: Procedure: Tetric N Ceram Bulkfill application
- Cention Forte (Active Comparator): Cention Forte was randomly applied to patients.
  Interventions: Procedure: Cention Forte application
- Stela Automix (Active Comparator): Stela automix was randomly applied to patients.
  Interventions: Procedure: Stela Automix
- Activa BioActive Restorative (Active Comparator): Activa BioActive Restorative was randomly applied to patients.
  Interventions: Procedure: Activa BioActive Restorative

INTERVENTIONS:
Procedure: Tetric N Ceram Bulkfill application — Selective enamel etching was performed with 37% phosphoric acid followed by a universal adhesive system application to all cavity surfaces and LED cured. The bulk-fill composite resin was placed in a single increment according to the manufacturer's recommendations and light-cured for 20 seconds. Excess material was removed using flame-shaped diamond finishing burs. Occlusion was assessed with articulation paper, and premature or undesirable contact points were adjusted as necessary.
  Arms: Tetric N-Ceram BulkFill
Procedure: Cention Forte application — A drop of Cention Primer was mixed in its wheel for 5 seconds and actively applied to the cavity for 10 seconds, followed by gentle air-drying. The Cention Forte capsule was then mixed for 15 seconds in a capsule mixer and placed in bulk into the prepared cavity using the manufacturer's delivery gun. Light curing was performed for 20 seconds with an LED unit (1300 mW/cm²; ZenoLite, President, Germany). Excess material was removed using flame-shaped diamond finishing burs. Occlusion was assessed with articulation paper, and any premature or undesirable contact points were adjusted accordingly. Final polishing was performed with OptraGloss polishing wheels (Ivoclar Vivadent) for 20 seconds.
  Arms: Cention Forte
Procedure: Stela Automix — Stela Primer was applied to the cavity surfaces and margins for 10 seconds. After a 5-second waiting period, the primer was gently air-dried for 2-3 seconds. The Stela Automix injector tip was then angled as needed and inserted into the cavity to deliver the material. The restoration was allowed to self-cure for 4 minutes. Occlusion was evaluated using articulation paper, and any premature or undesired contact points were adjusted as necessary. Final polishing was performed with OptraGloss polishing wheels (Ivoclar Vivadent) for 20 seconds.
  Arms: Stela Automix
Procedure: Activa BioActive Restorative — Selective enamel etching was performed with 37% phosphoric acid for 15 seconds, followed by thorough rinsing and air-drying. A universal adhesive system (Tetric N-Bond Universal, Ivoclar Vivadent) was applied to all cavity surfaces, including enamel, for 20 seconds, air-thinned, and light-cured for 20 seconds using an LED unit (1300 mW/cm²; ZenoLite, President, Germany). Following the manufacturer's instructions, the placement tip was inserted into the cavity using the dedicated placement gun, and the material was delivered in bulk. Light curing was performed for 20 seconds. Excess material was removed using flame-shaped diamond finishing burs. Occlusion was assessed with articulation paper, and premature or undesirable contact points were adjusted as needed. Final polishing was performed with OptraGloss polishing wheels (Ivoclar Vivadent) for 20 seconds.
  Arms: Activa BioActive Restorative

SUMMARY:
The aim of this clinical study is to evaluate the performance of three different bioactive restorative materials against a composite resin for a period of 9 months.

This randomized, split-mouth, single-center trial was performed on patients having occlusal caries (ICDAS 3 and 4) in both molars of the same jaw. The restorative materials used were Tetric N-Ceram Bulk-fill (control, Ivoclar Vivadent, Liechtenstein), Stela (SDI, Australia), Cention Forte (Ivoclar) and Activa BioActive Restorative (Pulpdent, USA). The restorations were evaluated at baseline, 3-6 and 9-month according to FDI-2 criteria, in terms of functional, biological, and aesthetic parameters, by two experienced evaluators.

DETAILED DESCRIPTION:
Objectives: To clinically evaluate the performance of three different bioactive restorative materials against a composite resin for a period of 9 months.

Materials and Methods: This randomized, split-mouth, single-center trial was performed on patients having occlusal caries (ICDAS 3 and 4) in both molars of the same jaw. The restorative materials used were Tetric N-Ceram Bulk-fill (control, Ivoclar Vivadent, Liechtenstein), Stela (SDI, Australia), Cention Forte (Ivoclar) and Activa BioActive Restorative (Pulpdent, USA). The material allocation was randomly assigned by a drawing lot. The restorations were evaluated at baseline, 3-6 and 9-month according to FDI-2 criteria, in terms of functional, biological, and aesthetic parameters, by two experienced evaluators. Chi-square test was used to compare the variables in the categories. Mann-Whitney U test and paired T test compared the difference in scores for the groups (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 16 with permanent dentition
* Individuals with a total of four vital molar teeth requiring restoration (ICDAS 3-4), two on each side of the same jaw
* Individuals with posterior contact with antagonist teeth
* Individuals who are reliable, cooperative, and willing to participate in periodic follow-ups

Exclusion Criteria:

* Individuals whose antagonist teeth were missing or have crowns, bridges, etc.
* Individuals with history of alcohol, drug, or medication addiction.
* Individuals with pulp exposure during cavity preparation or a cavity depth exceeding 2-4 mm.
* Individuals known to be unable to attend follow-up appointments.
* Individuals with allergies to the products used in the procedure.
* Individuals with severe tooth grinding or bruxism.
* Individuals with caries conditions classified as ICDAS 5 and 6.
* Pregnant or breastfeeding individuals and individuals planning pregnancy during the study.

Ages: 20 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
FDI-2 evaluation criteria for functional properties | 2 years
  Clinical evaluations were conducted using the FDI-2 criteria by two experienced, calibrated, and blinded evaluators for functional properties (category F). fracture/displacement of the material, marginal adaptation, form and contour, occlusion, and wear) were scored. Scores of 1-3 indicate clinically acceptable and successful restorations, score 4 indicates clinically inadequate but repairable defects, and score 5 represents clinically unacceptable restorations.

SECONDARY OUTCOMES:
FDI-2 evaluation criteria for biological properties | 2 years
  Clinical evaluations were conducted using the FDI-2 criteria by two experienced, calibrated, and blinded evaluators for biological properties (category B). Secondary caries, integrity of tooth structure at restoration margins, post-operative sensitivity, and pulp status) were scored. Scores of 1-3 indicate clinically acceptable and successful restorations, score 4 indicates clinically inadequate but repairable defects, and score 5 represents clinically unacceptable restorations.

OTHER OUTCOMES:
FDI-2 evaluation criteria for aesthetic properties | 2 years
  Clinical evaluations were conducted using the FDI-2 criteria by two experienced, calibrated, and blinded evaluators for aesthetic properties (category A). Surface gloss and texture, margin staining, color matching, anatomical form were scored. Scores of 1-3 indicate clinically acceptable and successful restorations, score 4 indicates clinically inadequate but repairable defects, and score 5 represents clinically unacceptable restorations.

CONTACTS AND LOCATIONS:
Overall Officials: Cankut Canevi, DDS, Principal Investigator — Ege University School of Dentistry Department of Restorative Dentistry
Locations (1):
- Ege University School of Dentistry, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No